CLINICAL TRIAL: NCT05777655
Title: Improving Adherence to Statin Therapy Through a Medication Management Application (STAPP)
Brief Title: Improving Adherence to Statin Therapy Through a Medication Management Application
Acronym: STAPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Benedikt Frank, Assistant Professor (PD) Dr. med, University Hospital, Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21-10444
Record Dates: First submitted 2023-02-22; First posted 2023-03-21 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Atherosclerosis
Keywords: Smartphone Application; Medication Therapy Management
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medication management app (Experimental): Standard of care (statin prescription, targeted monitoring of individual LDL-C values by primary care physician) + medication management app and follow-up visits at our institution at 6 and 18 months
  Interventions: Other: Medication management app (mediteo m+, Mediteo GmbH, Heidelberg)
- Standard of care (No Intervention): Statin prescription, targeted monitoring of individual LDL-C values by primary care physician and follow-up visits at our institution at 6 and 18 months

INTERVENTIONS:
Other: Medication management app (mediteo m+, Mediteo GmbH, Heidelberg) — Free access to a study version of the medication management app mediteo m+ for reminders and documentation of statin therapy in addition to usual care
  Arms: Medication management app

SUMMARY:
Interventional study to compare standard of care vs standard of care plus the use of a medication therapy management smartphone app (mediteo m+, Mediteo GmbH, Heidelberg) in patients with atherosclerotic cardiovascular disease and indication to start high intensity statin therapy.

DETAILED DESCRIPTION:
Patients with atherosclerotic cardiovascular disease and indication to start high intensity statin therapy will be recruited during hospital-stay or in the neurovascular outpatient clinic of the Neurology Department as well as in the Department of Cardiology and Vascular Medicine at the University Hospital Essen. Participants will be randomly allocated 1:1 to the intervention or control arm and all will receive a Low density Lipoprotein-Cholesterin (LDL-C) target and a statin-prescription as standard of care. All patients will be asked to take the prescribed statin in the evening and to provide LDL-C values measured by the family physician after 6 and 18 months. Additional blood will be collected after 6 and 18 months to control for cardiovascular risk-factors in the study center (LDL-C amongst others). In addition, the intervention group will receive free access to a study version of the medication management app mediteo m+ (Mediteo GmbH, Heidelberg). Installation of the app will be performed on the day of enrolment. After entering the medication, the app will remind the patient to take his or her statin therapy according to the therapy plan. Each intake has to be confirmed by the patient, either directly via the reminder notification or in the app. In addition, the app can be used to set reminders to go the family physician to take LDL-C values and to document the personal LDL-C values. The endpoint assessment will be performed in blinded manner.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Atherosclerosis (neurovascular, cardiac or peripheral) with an indication to start a high intensity statin-therapy (equivalent to 40mg of atorvastatin or 20mg of rosuvastatin; start of statin therapy +/- 10 days of enrolment)
* Statin naivety
* LDL-C >100 mg/dl. No older than 21 days

Exclusion Criteria:

* Inability to take medication independently or to use the mediteo m+ app independently (e.g. people in need of care, people with dementia)
* Patient has no own smartphone (no device provided for this study)
* Prior drug therapy to lower LDL-C within the last 30 days
* Active cancer (defined as a diagnosis of cancer within 6 months before enrolment, any treatment for cancer within the previous 6 months, or recurrent or metastatic cancer) or other severe concomitant disease with a life expectancy of <6 months
* Use of a digital therapy management application (including mediteo or mediteo m+) within the last month
* Participation in another interventional trial
* Pregnancy
* Inability or unwillingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Relative change in LDL-C | 6 months
  Relative change in LDL-C (mg/dl) after 6 months measured by study site (or according to the value measured by the family physician, if the value measured by the study site is not available after 6 months) as compared to baseline-value

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS)-Score after 6 months | 6 months
  Change in mRS [0 to 6, higher scores indicating worse outcome] after 6 months
Proportion of available LDL-C values measured by the family physician after 6 months | 6 months
  Proportion of available LDL-C values measured by the family physician after 6 months
Relative change in high density lipoprotein-cholesterol (HDL-C) after 6 months | 6 months
  Relative change in HDL-C (mg/dl) after 6 months as compared to baseline-value
Relative change in total cholesterol after 6 months | 6 months
  Relative change in total cholesterol (mg/dl) after 6 months as compared to baseline-value
Relative change in hemoglobin A1C (HbA1c) after 6 months | 6 months
  Relative change in HbA1c (%) after 6 months as compared to baseline-value
Relative change in high-sensitivity C-reactive protein (hsCRP) after 6 months | 6 months
  Relative change in hsCRP (mg/dl) after 6 months as compared to baseline-value
Relative change in Lipoprotein (a) after 6 months | 6 months
  Relative change in Lipoprotein (a) (mg/dl) after 6 months as compared to baseline-value
Relative change in glutamic oxaloacetic transaminase (GOT) after 6 months | 6 months
  Relative change in GOT (U/l) after 6 months as compared to baseline-value
Relative change in glutamate-pyruvate transaminase (GPT) | 6 months
  Relative change in GPT (U/l) after 6 months as compared to baseline-value
Relative change in creatine kinase (CK) after 6 months | 6 months
  Relative change in CK (U/l) after 6 months as compared to baseline-value
Adherence to statin therapy as measured by the German version of the Medication Adherence Report Scale (MARS-D) after 6 months | 6 months
  Adherence to statin therapy after 6 months as measured by the German version of the Medication Adherence Report Scale as measured by MARS-D, range 5-25, higher scores indicating better adherence
Adherence to statin therapy as measured by the German version of the A14 scale after 6 months | 6 months
  Measured by the German version of the A14 scale, range 0 - 56, lower scores indicating better adherence
Change in Quality of life score EQ-5D-5L after 6 months | 6 months
  Change in Quality of life score EQ-5D-5L is a standardised measure of health status developed by the EuroQol Group including 5 dimensions, 5 levels and the EQ visual analogue scale [VAS] from 0 to 100 with higher values indicating higher quality of life
Change in Beliefs about Medicines Questionnaire (BMQ) after 6 months | 6 months
  The BMQ consists of two sections assessing personal beliefs about the necessity of prescribed medication (5 items) and concerns (5 items). Scores range from 5 to 25 with higher scores indicating a higher degree of necessity/concern.
Incidence of major vascular events after 6 months | 6 months
  Incidence of cardiovascular death, myocardial infarction, stroke, hospitalization for unstable angina or urgent coronary revascularization therapy after 6 months
Change in highest degree of extracranial stenosis after 6 months | 6 months
  Change in highest degree of extracranial stenosis (%) as determined by carotid ultrasound using North American Carotid Endarterectomy Trial (NASCET) criteria after 6 months
Change in maximum height of largest carotid plaque after 6 months | 6 months
  Change in maximum height of largest carotid plaque (mm) on carotid ultrasound after 6 months
Change in longitudinal area of largest carotid plaque after 6 months | 6 months
  Change in longitudinal area of largest carotid plaque [mm2] on carotid ultrasound after 6 months
Change in cross-sectional area of largest carotid plaque after 6 months | 6 months
  Change in cross-sectional area of largest carotid plaque [mm2] on carotid ultrasound after 6 months
Relative change in LDL-C after 18 months | 18 months
  Relative change in LDL-C (mg/dl) after 18 months measured by study site (or according to the value measured by the family physician, if the value measured by the study site is not available) as compared to baseline-value
Modified Rankin Scale (mRS)-Score after 18 months | 18 months
  Change in mRS [0 to 6, higher scores indicating worse outcome] after 18 months
Proportion of available LDL-C values measured by the family physician after 18 months | 18 months
  Proportion of available LDL-C values measured by the family physician after 18 months
Relative change in high density lipoprotein-cholesterol (HDL-C) after 18 months | 18 months
  Relative change in HDL-C (mg/dl) after 18 months as compared to baseline-value
Relative change in total cholesterol after 18 months | 18 months
  Relative change in total cholesterol (mg/dl) after 18 months as compared to baseline-value
Relative change in hemoglobin A1C (HbA1c) after 18 months | 18 months
  Relative change in HbA1c (%) after 18 months as compared to baseline-value
Relative change in high-sensitivity C-reactive protein (hsCRP) after 18 months | 18 months
  Relative change in hsCRP (mg/dl) after 18 months as compared to baseline-value
Relative change in Lipoprotein (a) after 18 months | 18 months
  Relative change in Lipoprotein (a) (mg/dl) after 18 months as compared to baseline-value
Relative change in glutamic oxaloacetic transaminase (GOT) after 18 months | 18 months
  Relative change in GOT (U/l) after 18 months as compared to baseline-value
Relative change in glutamate-pyruvate transaminase (GPT) after 18 months | 18 months
  Relative change in GPT (U/l) after18 months as compared to baseline-value
Relative change in creatine kinase (CK) after 18 months | 18 months
  Relative change in CK (U/l) after 18 months as compared to baseline-value
Adherence to statin therapy as measured by the German version of the Medication Adherence Report Scale (MARS-D) after 18 months | 18 months
  Adherence to statin therapy after 18 months as measured by the German version of the Medication Adherence Report Scale as measured by MARS-D, range 5-25, higher scores indicating better adherence
Adherence to statin therapy as measured by the German version of the A14 scale after 18 months | 18 months
  Measured by the German version of the A14 scale, range 0 - 56, lower scores indicating better adherence
Change in Quality of life score EQ-5D-5L after 18 months | 18 months
  Change in Quality of life score EQ-5D-5L is a standardised measure of health status developed by the EuroQol Group including 5 dimensions, 5 levels and the EQ visual analogue scale [VAS] from 0 to 100 with higher values indicating higher quality of life
Change in Beliefs about Medicines Questionnaire (BMQ) after 18 months | 18 months
  The BMQ consists of two sections assessing personal beliefs about the necessity of prescribed medication (5 items) and concerns (5 items). Scores range from 5 to 25 with higher scores indicating a higher degree of necessity/concern.
Incidence of major vascular events after 18 months | 18 months
  Incidence of cardiovascular death, myocardial infarction, stroke, hospitalization for unstable angina or urgent coronary revascularization therapy after 18 months
Change in highest degree of extracranial stenosis after 18 months | 18 months
  Change in highest degree of extracranial stenosis (%) as determined by carotid ultrasound using North American Carotid Endarterectomy Trial (NASCET) criteria after 18 months
Change in maximum height of largest carotid plaque after 18 months | 18 months
  Change in maximum height of largest carotid plaque (mm) on carotid ultrasound after 18 months
Change in longitudinal area of largest carotid plaque after 18 months | 18 months
  Change in longitudinal area of largest carotid plaque [mm2] on carotid ultrasound after 18 months
Change in cross-sectional area of largest carotid plaque after 18 months | 18 months
  Change in cross-sectional area of largest carotid plaque [mm2] on carotid ultrasound after 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No